CLINICAL TRIAL: NCT04842292
Title: Utilization of Nebulized Heparin for Patients Receiving Mechanical Ventilation for COVID19-associated Acute Respiratory Failure
Brief Title: Nebulized Heparin for COVID19-associated Acute Respiratory Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Brittany Bissell (Other)
Responsible Party: Sponsor-Investigator, Brittany Bissell, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65139
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Heparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized heparin (Experimental): Nebulized heparin 25,000 units in 3 mL inhalation every 6 hours
  Interventions: Drug: Heparin
- Nebulized placebo (Placebo Comparator): Sodium chloride 0.9% 5 mL inhalation every 6 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Heparin — Nebulized heparin 25,000 units every 6 hours
  Arms: Nebulized heparin
Drug: Placebo — Sodium chloride 0.9% every 6 hours
  Arms: Nebulized placebo

SUMMARY:
The objective of the current study is to investigate the utilization of nebulized heparin to circumvent pathologic changes in COVID-19 and prevent harmful effects possible with systemic anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted with confirmed COVID-19 receiving mechanical ventilation for ARDS (paO2/FiO2 ratio =300) within 48 hours

Exclusion Criteria:

* Allergy to heparin
* Any history of heparin-induced thrombocytopenia
* High risk of bleeding (platelet count < 50,000/µL or international normalized ratio > 1.5)
* Patients with known bleeding disorders (i.e. hemophilia or von Willebrand Disease)
* Active bleeding
* Pulmonary bleeding during this hospital admission (Pulmonary bleeding is frank bleeding in the lungs, trachea or bronchi with repeated hemoptysis, or requiring repeated suctioning, and temporally associated with acute deterioration in respiratory status)
* Neurosurgical procedures during this hospital admission or such procedures are planned
* Epidural catheter in place
* Any history of intracranial, spinal or epidural hemorrhage
* Tracheostomy in place
* Cervical spinal cord injury associated with reduced long-term ability to breathe independently
* Spinal or peripheral nerve disease with a likely prolonged reduction in the ability to breathe independently
* Receiving extra-corporeal membrane oxygenation or continuous renal replacement therapy
* Usually treated with hemodialysis or peritoneal dialysis for end-stage renal failure
* Death is deemed imminent or inevitable or there is an underlying disease with a life expectancy of fewer than 90 days
* Pregnant or might be pregnant.
* Objection from the treating clinician
* Consent refused by the patient or substitute decision maker.
* History of thrombosis (VTE or cardiovascular event)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany D Bissell, Principal Investigator — University of Kentucky
Locations (1):
- UK Healthcare, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants were enrolled. To protect privacy, data will not be presented for each arm.
Groups:
- Participants: Two participants were enrolled in this study. Due to the possibility that participants could reasonably be identified due to low enrollment, data for the two arms will be combined.
Period: Overall Study
Arm/Group | Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Two participants were enrolled.
Arm/Group | Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean PaO2/FiO2 Ratio
Time Frame: Within the first 10 days of ICU stay or up until ICU discharge, whichever occurs first
Population: Two participants were enrolled in this study. Due to the possibility that participants could reasonably be identified due to low enrollment, data cannot be presented.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Participants: Two participants were enrolled in this study. Due to the possibility that participants could reasonably be identified due to low enrollment, data cannot be presented.
Arm/Group | Participants
Number analyzed (Participants) | 2
units on a scale | NA (NA) — Due to the possibility that individual participant data could be identified since there were only 2 participants, data cannot be presented without risking participant privacy.

2. Secondary Outcome: Clinically Significant Bleeding
Time Frame: Up to discharge or 3 months following enrollment, whichever occurs first
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants
Number analyzed (Participants) | 2
units on a scale | NA (NA) — Due to the possibility that individual participant data could be identified since there were only 2 participants, data cannot be presented without risking participant privacy.

3. Secondary Outcome: Incidence of Venous Thromboembolism
Time Frame: Up to discharge or 3 months following enrollment, whichever occurs first
Population: as for outcome 1
Measure: Number; unit: Incidence
Arm/Group | Participants
Number analyzed (Participants) | 2
Incidence | NA — Due to the possibility that individual participant data could be identified since there were only 2 participants, data cannot be presented without risking participant privacy.

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT04842292/Prot_ICF_000.pdf